CLINICAL TRIAL: NCT00699153
Title: Safety and Efficacy of Loteprednol Etabonate in an Ophthalmic Base vs Vehicle for the Treatment of Inflammation Following Cataract Surgery
Brief Title: Loteprednol Etabonate in an Ophthalmic Base vs Vehicle for the Treatment of Inflammation Following Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 526
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Results first posted 2010-09-23 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Ocular Inflammation
MeSH Terms: interventions — Loteprednol Etabonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Loteprednol Etabonate (Experimental): Loteprednol Etabonate 0.5%
  Interventions: Drug: Loteprednol Etabonate
- Vehicle (Placebo Comparator): Vehicle of Ophthalmic Loteprednol Etabonate
  Interventions: Drug: Vehicle of Ophthalmic Loteprednol Etabonate

INTERVENTIONS:
Drug: Loteprednol Etabonate — Loteprednol Etabonate in an ophthalmic base will be administered to study eye 4 times a day(QID) for 14 days.
  Arms: Loteprednol Etabonate
Drug: Vehicle of Ophthalmic Loteprednol Etabonate — Vehicle of ophthalmic loteprednol etabonate administered postoperatively to study eye 4 times a day(QID) for 14 days.
  Arms: Vehicle

SUMMARY:
Evaluation of the clinical safety and efficacy of loteprednol etabonate in an ophthalmic base, when compared to vehicle for the treatment of inflammation following cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects at least 18 years of age
* Subjects who have the ability to understand and sign an informed consent form and provide Health Insurance Portability and Accountability Act (HIPAA) authorization.
* Subjects who are candidate for routine, uncomplicated cataract surgery.
* Subjects who are not of childbearing potential or subjects who have a negative urine pregnancy test result at screening.
* Subjects must be willing and able to comply with all treatment and follow- up procedures.

Exclusion Criteria:

* Subjects who have known hypersensitivity or contraindication to the study drug or its components.
* Subjects who have a history or presence of chronic generalized systemic disease that the investigator feels might increase the risk to the subject or compound the result of the study.
* Subjects who have a severe/serious ocular condition, or any other unstable medical condition that, in the Investigator's opinion, may preclude study treatment or follow-up.
* Subjects with elevated intraocular pressure (>/= 21 mm Hg), uncontrolled glaucoma, or being treated for glaucoma in the study eye.
* Subjects who are monocular or have pinholed Snellen VA 20/200 or worse in the non-study eye.
* Subjects who have had ocular surgery in the study eye within 3 months or in the fellow eye within 2 weeks prior to the screening visit.
* Women who are pregnant or breast feeding.
* Subjects who have participated in an investigational drug or device study within the last 30 days.
* Subjects previously randomized in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2008-06; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Trusso, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Cornerstone Eye Wear, High Point, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 16 sites in the US. The first participant was enrolled June 20, 2008 and the last participant visit was May 1, 2009.
Pre-assignment Details: 405 participants, who were candidates for routine, uncomplicated cataract surgery were enrolled in the study.
Groups:
- Loteprednol Etabonate: Loteprednol Etabonate Ophthalmic Ointment 0.5%
Period: Overall Study
Arm/Group | Loteprednol Etabonate | Vehicle
Started | 203 (Intent to treat population) | 202 (Intent to treat population)
Completed | 200 | 200
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 0 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Travel Problem | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Loteprednol Etabonate | Vehicle | Total
Number analyzed (Participants) | 203 | 202 | 405
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (9.13) | 69.2 (9.36) | 68.8 (9.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 115 | 230
  Male | 88 | 87 | 175
Race/Ethnicity, Customized [Number; unit: participants]
  White | 182 | 178 | 360
  Black/African American | 13 | 16 | 29
  American Indian/Alaskan Native | 2 | 0 | 2
  Asian | 5 | 6 | 11
  Native Hawiian/Pacific Islander | 0 | 1 | 1
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Participants With Complete Resolution of Anterior Chamber Cells and Flare. Grade=0
Description: A combination of the grades for inflammatory cells and flare in the anterior chamber. Cells: accumulation of white blood cells in aqueous. 0=No cells seen; 1=1-5 cells; 2=6-15 cells; 3=16-30 cells; 4= >30 cells. Flare: Scattering of a slit lamp light beam when directed into the anterior chamber (Tyndall effect). 0=None; 1=Mild; 2=Moderate; 3=Severe; 4=Very severe.
Time Frame: Postoperative day 8 (Visit 5)
Population: Intent to treat population, subjects who had missing data or took rescue medication prior to visit 5 were imputed as no.
Measure: Number; unit: participants
Arm/Group | Loteprednol Etabonate | Vehicle
Number analyzed (Participants) | 203 | 202
participants | 64 | 23

2. Primary Outcome: Participants With Grade 0 (no) Pain
Description: Pain: A positive sensation of the eye, including foreign body sensation, stabbing, throbbing, or aching. Grade 0 = None; 1=Minimal; 2=Mild; 3=Moderate; 4=Moderately Severe; 5=Severe
Time Frame: Postoperative day 8 (Visit 5)
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Loteprednol Etabonate | Vehicle
Number analyzed (Participants) | 203 | 202
participants | 149 | 83

3. Secondary Outcome: Participants With Complete Resolution of Anterior Chamber Cells and Flare, at Each Visit.
Description: as for outcome 1
Time Frame: At each visit: Visit 4-7, postoperative days 3-18
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Loteprednol Etabonate | Vehicle
Number analyzed (Participants) | 203 | 202
participants
  Visit 4, postoperative day 3 | 10 | 9
  Visit 5, postoperative day 8 | 64 | 23
  Visit 6, posoperative day 15 | 107 | 42
  Visit 7, postoperative day 18 | 100 | 46

4. Secondary Outcome: Mean Change From Baseline to Each Follow-up Visit in Anterior Chamber Cells and Flare
Description: as for outcome 1
Time Frame: Postoperative Day 3-18 (Each follow-up Visit 4-7)
Population: Intent to treat population.
Measure: Mean (Standard Deviation); unit: Composite scores
Arm/Group | Loteprednol Etabonate | Vehicle
Number analyzed (Participants) | 203 | 202
Composite scores
  Visit 4, postoperative day 3 | -1.2 (1.20) | -0.6 (1.48)
  Visit 5, postoperative day 8 | -2.2 (1.51) | -0.8 (1.81)
  Visit 6, postoperative day 15 | -2.7 (1.58) | -1.1 (1.94)
  Visit 7, postoperative day 18 | -2.6 (1.59) | -1.1 (2.01)

ADVERSE EVENTS:
Time Frame: Following drug administration visit 3 (postoperative day 1) through visit 7 (postoperative day 18).
Description: Ocular treatment related ocular AE's in >/= 5% of Study Eyes, Either Treatment Group, Prior to Rescue Medication Use - Safety Population 204 Loteptednol, 201 Vehicle.
Arm/Group | Loteprednol Etabonate | Vehicle
Serious Adverse Events (participants affected / at risk) | 2/204 | 4/201
Other Adverse Events (participants affected / at risk) | 81/204 | 151/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Loteprednol Etabonate (N=204) | Vehicle (N=201)
Blocked arteries (Cardiac disorders) | 2 (2) | 2 (2) — One subject had 2 events of blocked arteries
Diabetic foot ulcer (Endocrine disorders) | 1 (1) | 1 (1)
Fall/Hip fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Pituitary tumor (Endocrine disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Loteprednol Etabonate (N=204) | Vehicle (N=201)
Anterior chamber inflammation (Eye disorders) | 49 (119) | 94 (241) — Ocular TEAEs Related to Study Drug in Study Eyes, Either Treatment Group, Prior to Rescue Medication Use - Safety Population
Eye Pain (Eye disorders) | 7 (119) | 17 (241) — Ocular TEAEs >/= 5% in Study Eyes, Either Treatment Group, Prior to Rescue Medication Use - Safety Population
Corneal Edema (Eye disorders) | 10 (119) | 12 (241) — Ocular TEAEs in >/= 5% of Study Eyes, Either Treatment Group, Prior to Rescue Medication Use - Safety Population
Conjunctival Hyperemia (Eye disorders) | 6 (119) | 15 (241) — Ocular TEAEs in >/= 5% of Study Eyes, Either Treatment Group, Prior to Rescue Medication Use - Safety Population
Ciliary Hyperemia (Eye disorders) | 5 (119) | 13 (241) — Ocular TEAEs in >/= 5% of Study Eyes, Either Treatment Group, Prior to Rescue Medication Use - Safety Population
Photophobia (Eye disorders) | 5 (119) | 12 (241) — Ocular TEAEs in >/= 5% of Study Eyes, Either Treatment Group, Prior to Rescue Medication Use - Safety Population
Iritis (Eye disorders) | 4 (119) | 12 (241) — Ocular TEAEs in >/= 5% of Study Eyes, Either Treatment Group, Prior to Rescue Medication Use - Safety Population
Uveitis (Eye disorders) | 4 (119) | 10 (241) — Ocular TEAEs in >/= 5% of Study Eyes, Either Treatment Group, Prior to Rescue Medication Use - Safety Population

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with, the Sponsor and such that confidential or proprietary information is not disclosed. Prior to publication or presentation, a copy of the final text should be forwarded by the Investigator(s) to the Sponsor or its designee for comment.